CLINICAL TRIAL: NCT06438042
Title: Prevention of Pressure Ulcers in Patients at High Risk of Developping Pressure Ulcers Using the Low-pressure Motorized Air Support Mattress With XTECH®25 Control Unit
Status: Recruiting | Type: Observational
Sponsor: SYSTAM (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A01556-39
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Pressure Ulcer
Keywords: Prevention; Pressure ulcer; Low air pressure motorised mattress
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in nursing homes or long-stay geriatrics department
  Interventions: Device: Use of a powered low air pressure motorised therapeutic mattress that combines the motorised and static technologies

INTERVENTIONS:
Device: Use of a powered low air pressure motorised therapeutic mattress that combines the motorised and static technologies — Patients with a high risk of pressure injury, without pressure injury, lying more than 20 hours a day, will ly a on a XTECH®25 mattress

SUMMARY:
The aim of the study is to determine the clinical value of using a a low air pressure motorised therapeutic mattress in the prevention of pressure injury (PI) in patients at medium to high risk.

This study is noncomparative, observational study.

Patients older than 18 years of age, with a high risk of PI, without PI, lying more than 20 hours a day on a XTECH®25 mattress will be included. The study will be conducted in nursing homes, and in long-stay geriatrics department.

Patients are followed up for 35 days. The use of the XTECH®25 mattress is associated with the usual PI prevention measures. The primary outcome is the percentage of patients who developed between day 0 and day 35 at least one PI of at least stage 2 on the sacrum, spine, or heel. Secondary endpoints are patient assessments of comfort, caregiver satisfaction, mattress noise level, and mattress safety.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with high risk of developing pressure ulcers (clinical judgment and a score <= 12 on the Braden scale (6 (maximum risk) to 23 (no risk))
* Patient without pressure injury on the day of inclusion
* Patient up lying more than 20 hours a day on XTECH®25 mattress
* Patient with a weight < 200 kg
* Patient (or a trusted third party) having been informed of the study and agreeing to participate

Exclusion Criteria:

* Patient at end of life (estimated life expectancy less than 6 months)
* Patient discharge from the establishment expected within two months
* Participants will be excluded from the study if they meet the following combination of criteria indicative of malnutrition according to the 2021 Haute Autorité de la Santé guidelines (Participants must meet at least one phenotypic criterion and one etiological criterion to be considered malnourished and therefore ineligible for inclusion in the study) :

A) One or more of the following phenotypic criteria:

1. Significant unintentional weight loss: A weight loss of ≥ 5% within 1 month or ≥ 10% within 6 months
2. Low Body Mass Index (BMI): BMI < 18.5 kg/m² for individuals under 70 years old, BMI < 21 kg/m² for individuals aged 70 years and older
3. Reduced Muscle Mass
4. Evident reduction in muscle mass AND

B) One of the following etiological criteria:

1. Inadequate nutritional intake:
2. Nutritional intake less than 50% of the energy requirements for more than one week
3. Reduced food intake for more than two weeks
4. Presence of Disease or Stress Metabolism
5. Acute or chronic illness, or any condition causing metabolic stress that increases energy requirements .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in nursing homes or long-stay geriatrics department
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who developed at least one stage 2 pressure injury | 35 days after installation on the mattress (at day 35)
  Percentage of patients who developed at least one stage 2 PI of the sacrum, backbone, or heel (areas of support when lying down)

SECONDARY OUTCOMES:
Percentage of patients who developed a o pressure injury (any stage), other than those of the sacrum, backbone, or heel between | 35 days after installation on the mattress (at day 35)
Assessment by the patient (or family or staff in the case of incapacity) of the comfort of the mattress (general comfort, stability) | 35 days after installation on the mattress (at day 35)
  On a scale from 0 (not satisfied at all) to 4 (very satisfied)
Assessment by the nursing staff with the use of the mattress (implementation, cleaning maintenance turning, changing to a sitting position) | 35 days after installation on the mattress (at day 35)
  On a scale from 0 (not satisfied at all) to 4 (very satisfied)
Assessment of the degree of maceration | On a scale from 1 (constantly moist) to 4 rarely moist
  On a scale from 1 (constantly moist) to 4 rarely moist
Assessment of mattress safety | At day 35
  By collecting any adverse event or mattress malfunction during the follow up

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie MEAUME, Principal Investigator — Hôpital ROSCHILD
Locations (1):
- Multiples locations, Multiple Locations, France